CLINICAL TRIAL: NCT03204344
Title: Impact of Preoperative Oral Carbohydrate on Recovery in Diabetic Patients After Gastrointestinal Surgery: a Pilot Randomized Controlled Trial
Brief Title: Preoperative Oral Carbohydrate and Postoperative Recovery in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-Xin Wang (Other)
Responsible Party: Sponsor-Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017[1362]
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Surgery
Keywords: Gastrointestinal surgery; Preoperative oral carbohydrate; Diabetic patients; Postoperative recovery
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: This is a outcomes assessor-blinded, randomized controlled trial with two parallel arms.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor who perform postoperative follow-up is masked to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): For all patients, 2 bottles of oral carbohydrate (Outfast, 710 ml) is provided between 22:00-24:00 on the day before surgery. Subcutaneous insulin is administered before drinking.
  For patients who entered operating room before 12:00, 1 bottle of oral carbohydrate (Outfast) is provided at 6:00 on the day of surgery. For patients who enter the operating room after 12:00, another bottle of oral carbohydrate (Outfast) is provided at least 2 hours before entering the operating room. Subcutaneous insulin is administered before drinking.
  Interventions: Dietary Supplement: Oral carbohydrate (Outfast)
- Control group (Sham Comparator): For all patients, routine fasting (drinking water allowed) begins from 22:00 on the day before surgery， water fasting begins from 6:00 on the day of surgery.
  For patients who enter the operating room before 12:00, no oral or intravenoous fluid is provided from 6:00. For patients who enter the operating room after 12:00, 5% glucose (500-1000 ml) is provided by intravenous infusion from 6:00 on the day of surgery. Intravenous insulin is added (glucose:insulin=4-6:1). Electrolytes (such as sodium chloride, potasium chloride, magnesium sulfate) are added when becessary.
  Interventions: Other: Routine fasting

INTERVENTIONS:
Dietary Supplement: Oral carbohydrate (Outfast) — For all patients, 2 bottles of oral carbohydrate (Outfast, 710 ml) is provided between 22:00-24:00 on the day before surgery. Subcutaneous insulin is administered before drinking. The dose of insulin is calculated by an endocrinologist according to patients' daily glucose controlling plan.
  For patients who entered operating room before 12:00, 1 bottle of oral carbohydrate (Outfast) is provided at 6:00 on the day of surgery. For patients who enter the operating room after 12:00, another bottle of oral carbohydrate (Outfast) is provided at least 2 hours before entering the operating room. Subcutaneous insulin is administered before drinking. The dose of insulin is calculated is the same way as described above.
  Arms: Intervention group
Other: Routine fasting — For all patients, routine fasting (water drinking allowed) begin from 22:00 on the day before surgery until entering the operating room on the day of surgery.
  For patients who enter the operating room before 12:00, no oral or intravenoous fluid is provided. For patients who enter the operating room after 12:00, 5% glucose (500-1000 ml) is provided by intravenous infusion from 6:00 on the day of surgery. Intravenous insulin is added in the 5% glucose (glucose:insulin=4-6:1). Electrolytes (such as sodium chloride, potasium chloride, and magnesium sulfate) are added when considered necessary.
  Arms: Control group

SUMMARY:
For non-diabetic patients undergoing gastrointestinal surgery, preoperative oral carbohydrate improves postoperative recovery. The purpose of this pilot study is to investigate the impact of preoperative oral carbohydrate (outfast®) on the recovery in diabetic patients after gastrointestinal surgery.

DETAILED DESCRIPTION:
Studies show that avoiding long-time fasting by oral carbohydrates 2 hours before surgery attenuates discomfort and anxiety; it also reduces stress, insulin resistance and catabolism in patients undergoing gastrointestinal surgery, resulting in earlier recovery of gastrointestinal function and short length of hospital stay after surgery. However, for diabetic patients scheduled to undergo gastrointestinal surgery, the risks and benefits of preopertive oral carbohydrate remain unclear. The purpose of this pilot study is to investigate the impact of preoperative oral carbohydrate (outfast®) on the recovery in diabetic patients after gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years and beyond;
2. Diagnosed with type 2 diabetes before surgery;
3. Scheduled to undergo elective gastrointestinal surgery with anticipated duration of 2 hours or more;
4. Provide signed writen informed consents.

Exclusion Criteria:

1. Refuse to participate in the study;
2. Diagnosed with diaphragmatic hernia, gastric esophageal reflux disease or pregnancy;
3. Previous history of total or partial gastrectomy;
4. Preoperative New York Heart Assocition (NYHA) class IV, renal failure (requirement of renal replacement therapy), severe hepatic disease (Child-Pugh class C), or American Society of Anesthesiologists (ASA) class IV or higher;
5. Preoperative pyloric and/or intestinal obstruction;
6. Combined surgery on other intra-abdominal organs or other parts of the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Recovery of gastrointestinal function | From end of surgery until the time of first flatus and defecation, assessed up to 7 days after surgery.
  Time to first flatus and defecation after surgery.

SECONDARY OUTCOMES:
Subjective feelings | Before anesthesia induction and at 4-6 hours after surgery.
  Four subjective feelings, including the degree of being thirsty, hungry, tired and anxious, are assessed with Numeric Rating Scale (NRS, an 11-point scale where 0 = no feeling at all and 10 = the worst feeling).
Blood glucose variation | From 22:00 on the day before surgery until 24 hours after surgery.
  Difference between the highest and the lowest blood glucose levels.
Insulin resistance (in part of patients) | Assessed at 24 hours after surgery.
  Insulin resistance is calculated with the Homeostatic model assessment-insulin resistance (HOMA-IR) equation.
Length of stay in hospital after surgery. | From end of surgery until hospital discharge, up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of postoperative complications | From end of surgery until 30 days after surgery
  Postoperative complications are defined as newly occurred medical conditions that have harmful effects on patients' recovery and require therapeutic intervention.
Time to first walking in the ground and distance of walking after surgery. | During the first 5 days after surgery
  Time to first walking in the ground and distance of walking after surgery.
All cause 30-day mortality | At 30 days after surgery
  All cause 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available by contacting Dr. Xue Li (lixuepku@hotmail.com) after the trial is completed.

REFERENCES:
- [Background] Wang ZG, Wang Q, Wang WJ, Qin HL. Randomized clinical trial to compare the effects of preoperative oral carbohydrate versus placebo on insulin resistance after colorectal surgery. Br J Surg. 2010 Mar;97(3):317-27. doi: 10.1002/bjs.6963. PMID 20101593
- [Background] Hausel J, Nygren J, Thorell A, Lagerkranser M, Ljungqvist O. Randomized clinical trial of the effects of oral preoperative carbohydrates on postoperative nausea and vomiting after laparoscopic cholecystectomy. Br J Surg. 2005 Apr;92(4):415-21. doi: 10.1002/bjs.4901. PMID 15739210
- [Background] Singh BN, Dahiya D, Bagaria D, Saini V, Kaman L, Kaje V, Vagadiya A, Sarin S, Edwards R, Attri V, Jain K. Effects of preoperative carbohydrates drinks on immediate postoperative outcome after day care laparoscopic cholecystectomy. Surg Endosc. 2015 Nov;29(11):3267-72. doi: 10.1007/s00464-015-4071-7. Epub 2015 Jan 22. PMID 25609319
- [Background] Sada F, Krasniqi A, Hamza A, Gecaj-Gashi A, Bicaj B, Kavaja F. A randomized trial of preoperative oral carbohydrates in abdominal surgery. BMC Anesthesiol. 2014 Oct 17;14:93. doi: 10.1186/1471-2253-14-93. eCollection 2014. PMID 25364300
- [Background] Helminen H, Viitanen H, Sajanti J. Effect of preoperative intravenous carbohydrate loading on preoperative discomfort in elective surgery patients. Eur J Anaesthesiol. 2009 Feb;26(2):123-7. doi: 10.1097/EJA.0b013e328319be16. PMID 19142085
- [Background] Zelic M, Stimac D, Mendrila D, Tokmadzic VS, Fisic E, Uravic M, Sustic A. Influence of preoperative oral feeding on stress response after resection for colon cancer. Hepatogastroenterology. 2012 Jul-Aug;59(117):1385-9. doi: 10.5754/hge10556. PMID 22683955
- [Background] Zelic M, Stimac D, Mendrila D, Tokmadzic VS, Fisic E, Uravic M, Sustic A. Preoperative oral feeding reduces stress response after laparoscopic cholecystectomy. Hepatogastroenterology. 2013 Oct;60(127):1602-6. PMID 24634929
- [Background] Vigano J, Cereda E, Caccialanza R, Carini R, Cameletti B, Spampinato M, Dionigi P. Effects of preoperative oral carbohydrate supplementation on postoperative metabolic stress response of patients undergoing elective abdominal surgery. World J Surg. 2012 Aug;36(8):1738-43. doi: 10.1007/s00268-012-1590-4. PMID 22484570
- [Background] Lidder P, Thomas S, Fleming S, Hosie K, Shaw S, Lewis S. A randomized placebo controlled trial of preoperative carbohydrate drinks and early postoperative nutritional supplement drinks in colorectal surgery. Colorectal Dis. 2013 Jun;15(6):737-45. doi: 10.1111/codi.12130. PMID 23406311
- [Background] Perrone F, da-Silva-Filho AC, Adorno IF, Anabuki NT, Leal FS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, de Aguilar-Nascimento JE. Effects of preoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J. 2011 Jun 13;10:66. doi: 10.1186/1475-2891-10-66. PMID 21668975
- [Background] Faria MS, de Aguilar-Nascimento JE, Pimenta OS, Alvarenga LC Jr, Dock-Nascimento DB, Slhessarenko N. Preoperative fasting of 2 hours minimizes insulin resistance and organic response to trauma after video-cholecystectomy: a randomized, controlled, clinical trial. World J Surg. 2009 Jun;33(6):1158-64. doi: 10.1007/s00268-009-0010-x. PMID 19363695
- [Background] Makuuchi R, Sugisawa N, Kaji S, Hikage M, Tokunaga M, Tanizawa Y, Bando E, Kawamura T, Terashima M. Enhanced recovery after surgery for gastric cancer and an assessment of preoperative carbohydrate loading. Eur J Surg Oncol. 2017 Jan;43(1):210-217. doi: 10.1016/j.ejso.2016.07.140. Epub 2016 Aug 10. PMID 27554250
- [Background] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Background] Awad S, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of randomised controlled trials on preoperative oral carbohydrate treatment in elective surgery. Clin Nutr. 2013 Feb;32(1):34-44. doi: 10.1016/j.clnu.2012.10.011. Epub 2012 Nov 7. PMID 23200124
- [Background] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107
- [Background] An GQ, Zhao XL, Gao YC, Wang GY, Yu YM. [Effects of preoperative carbohydrate loading on the changes in serum tumor necrosis factor receptors 1 and 2 and insulin resistance in patients of colon carcinoma]. Zhonghua Yi Xue Za Zhi. 2008 Jul 29;88(29):2041-4. Chinese. PMID 19080431
- [Background] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Background] Alfonsi P, Slim K, Chauvin M, Mariani P, Faucheron JL, Fletcher D; Working Group of Societe francaise d'anesthesie et reanimation (SFAR); Societe francaise de chirurgie digestive (SFCD). French guidelines for enhanced recovery after elective colorectal surgery. J Visc Surg. 2014 Feb;151(1):65-79. doi: 10.1016/j.jviscsurg.2013.10.006. Epub 2013 Dec 27. PMID 24378143
- [Background] Horowitz M, O'Donovan D, Jones KL, Feinle C, Rayner CK, Samsom M. Gastric emptying in diabetes: clinical significance and treatment. Diabet Med. 2002 Mar;19(3):177-94. doi: 10.1046/j.1464-5491.2002.00658.x. PMID 11918620
- [Background] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374